CLINICAL TRIAL: NCT01780922
Title: Acute Bioavailability of Cranberry Polyphenols After A Single Dose In Healthy Adults and Its Antioxidative and Anti-Inflammatory Action
Brief Title: Effect of a Single Dose of Cranberry Beverage on Inflammation and Oxidative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: Ocean Spray Cranberries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 11369
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-06

CONDITIONS: Inflammation
Keywords: Inflammation; Oxidative Stress; Vaccinium macrocarpon
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Calorie Cranberry Juice Cocktail (Active Comparator): Beverage containing cranberry: one dose of 15.2 ounces consumed within 15 minutes
  Interventions: Other: Low Calorie Cranberry Juice Cocktail
- Cranberry Extract Beverage (Active Comparator): Beverage containing cranberry: one dose of 15.2 ounces consumed within 15 minutes
  Interventions: Other: Cranberry Extract Beverage
- Non-Cranberry Beverage (Placebo Comparator): Beverage absent cranberry: one dose of 15.2 ounces consumed within 15 minutes
  Interventions: Other: Non-Cranberry Beverage

INTERVENTIONS:
Other: Low Calorie Cranberry Juice Cocktail — Beverage containing cranberry at a dose of 15.2 ounces consumed within 15 minutes
  Arms: Low Calorie Cranberry Juice Cocktail
Other: Cranberry Extract Beverage — Beverage containing cranberry at a dose of 15.2 ounces consumed within 15 minutes
  Arms: Cranberry Extract Beverage
Other: Non-Cranberry Beverage — Beverage absent cranberry at a dose of 15.2 ounces consumed within 15 minutes
  Arms: Non-Cranberry Beverage

SUMMARY:
The purpose of this study is to determine the effects of a single dose of cranberry beverage in healthy adults on the kinetic uptake of polyphenol compounds and polyphenol metabolites, and antioxidative and anti-inflammatory activity.

DETAILED DESCRIPTION:
Participants will be randomized based on age, sex and BMI, and will consume a low-polyphenol diet 2 days prior to the intervention. On the day of the study, baseline blood and urine samples will be collected after an overnight fast. Participants will consume the assigned beverage within 15 minutes and blood collected at 2, 4, 8, and 24 h (10 mL/blood draw; total blood volume per period = 50 mL). Urine will be collected for polyphenol analysis during the following periods: 0-3, 3-6, 6-9, 9-12, 12-24 hours. After a one-week washout period, participants will receive their second and then the third beverage in a cross-over design; blood and urine sampling will be repeated at each of the 3 intervention periods.

ELIGIBILITY:
Inclusion Criteria:

* Men & women; aged 18-35 years
* BMI: 19-25 kg/m2

Exclusion Criteria:

* Any significant chronic disease, hypertension, ulcers, dyspepsia, lactose intolerance, allergy, psychotic illness
* Had major gastrointestinal surgery or on prescription or surgical treatment
* Any condition that may interfere with the digestion, absorption, metabolism or excretion of nutrients
* Regularly smoked in the previous 6 months
* On medication or ingested a prescribed drug at any time within the 14 days preceding study enrolment (excluding hormonal contraceptives and hormone replacement therapy) or over-the-counter preparation within 7 days preceding enrolment
* Risk factors for AIDS or known HIV positive status
* Pregnant or lactating
* High intake of chocolate or similar high polyphenol foods
* Regular intake of vitamin and polyphenol supplements
* Drug and alcohol misuse
* Currently participating or had participated in another clinical study during the previous 3 weeks
* Donated blood in the previous 3 weeks
* Exercise more than 3 times/week for longer than 45 min each time

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boon P Chew, PhD, Principal Investigator — Washington State University
Locations (1):
- WSU Bioactives Research Lab, Pullman, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- LCJC First, Then CLEB, Then Placebo: First Intervention (1 day) - Low Calorie Cranberry Juice Cocktail (LCJC): Beverage containing cranberry at a dose of 15.2 ounces consumed within 15 minutes Washout (7 days) Second Intervention (1 day) - Cranberry Leaf Extract Beverage (CLEB): Beverage containing cranberry at a dose of 15.2 ounces consumed within 15 minutes Washout (7 days) Third Intervention (1 day) - Placebo: Beverage absent cranberry at a dose of 15.2 ounces consumed within 15 minutes
- LCJC First, Then Placebo, Then CLEB: First Intervention (1 day) - Low Calorie Cranberry Juice Cocktail (LCJC): Beverage containing cranberry at a dose of 15.2 ounces consumed within 15 minutes Washout (7 days) Second Intervention (1 day) - Placebo: Beverage absent cranberry at a dose of 15.2 ounces consumed within 15 minutes Washout (7 days) Third Intervention (1 day) - Cranberry Leaf Extract Beverage (CLEB): Beverage containing cranberry at a dose of 15.2 ounces consumed within 15 minutes
- CLEB First, Then LCJC, Then Placebo: First Intervention (1 day) - Cranberry Leaf Extract Beverage (CLEB): Beverage containing cranberry at a dose of 15.2 ounces consumed within 15 minutes Washout (7 days) Second Intervention (1 day) - Low Calorie Cranberry Juice Cocktail (LCJC): Beverage containing cranberry at a dose of 15.2 ounces consumed within 15 minutes Washout (7 days) Third Intervention (1 day) - Placebo: Beverage absent cranberry at a dose of 15.2 ounces consumed within 15 minutes
- CLEB First, Then Placebo, Then LCJC: First Intervention (1 day) - Cranberry Leaf Extract Beverage (CLEB): Beverage containing cranberry at a dose of 15.2 ounces consumed within 15 minutes Washout (7 days) Second Intervention (1 day) - Placebo: Beverage absent cranberry at a dose of 15.2 ounces consumed within 15 minutes Washout (7 days) Third Intervention (1 day) - Low Calorie Cranberry Juice Cocktail (LCJC): Beverage containing cranberry at a dose of 15.2 ounces consumed within 15 minutes
- Placebo First, Then LCJC, Then CLEB: First Intervention (1 day) - Placebo: Beverage absent cranberry at a dose of 15.2 ounces consumed within 15 minutes Washout (7 days) Second Intervention (1 day) - Low Calorie Cranberry Juice Cocktail (LCJC): Beverage containing cranberry at a dose of 15.2 ounces consumed within 15 minutes Washout (7 days) Third Intervention (1 day) - Cranberry Leaf Extract Beverage (CLEB): Beverage containing cranberry at a dose of 15.2 ounces consumed within 15 minutes
- Placebo First, Then CLEB, Then LCJC: First Intervention (1 day) - Placebo: Beverage absent cranberry at a dose of 15.2 ounces consumed within 15 minutes Washout (7 days) Second Intervention (1 day) - Cranberry Leaf Extract Beverage (CLEB): Beverage containing cranberry at a dose of 15.2 ounces consumed within 15 minutes Washout (7 days) Third Intervention (1 day) - Low Calorie Cranberry Juice Cocktail (LCJC): Beverage containing cranberry at a dose of 15.2 ounces consumed within 15 minutes
Period: First Intervention (1 Day)
Arm/Group | LCJC First, Then CLEB, Then Placebo | LCJC First, Then Placebo, Then CLEB | CLEB First, Then LCJC, Then Placebo | CLEB First, Then Placebo, Then LCJC | Placebo First, Then LCJC, Then CLEB | Placebo First, Then CLEB, Then LCJC
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (7 Days)
Arm/Group | LCJC First, Then CLEB, Then Placebo | LCJC First, Then Placebo, Then CLEB | CLEB First, Then LCJC, Then Placebo | CLEB First, Then Placebo, Then LCJC | Placebo First, Then LCJC, Then CLEB | Placebo First, Then CLEB, Then LCJC
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | LCJC First, Then CLEB, Then Placebo | LCJC First, Then Placebo, Then CLEB | CLEB First, Then LCJC, Then Placebo | CLEB First, Then Placebo, Then LCJC | Placebo First, Then LCJC, Then CLEB | Placebo First, Then CLEB, Then LCJC
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (7 Days)
Arm/Group | LCJC First, Then CLEB, Then Placebo | LCJC First, Then Placebo, Then CLEB | CLEB First, Then LCJC, Then Placebo | CLEB First, Then Placebo, Then LCJC | Placebo First, Then LCJC, Then CLEB | Placebo First, Then CLEB, Then LCJC
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | LCJC First, Then CLEB, Then Placebo | LCJC First, Then Placebo, Then CLEB | CLEB First, Then LCJC, Then Placebo | CLEB First, Then Placebo, Then LCJC | Placebo First, Then LCJC, Then CLEB | Placebo First, Then CLEB, Then LCJC
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants: all participants received all interventions
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.7 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Reduced Glutathione (GSH) Concentrations in Red Blood Cells
Time Frame: 0, 2, 4, 8, 24 h
Measure: Mean (Standard Error); unit: mmol/L
Groups:
- Cranberry Leaf Extract Beverage: Beverage containing cranberry leaf extract: one dose of 15.2 ounces consumed within 15 minutes
  Cranberry Leaf Extract Beverage: Beverage containing cranberry at a dose of 15.2 ounces consumed within 15 minutes
Arm/Group | Low Calorie Cranberry Juice Cocktail | Cranberry Leaf Extract Beverage | Non-Cranberry Beverage
Number analyzed (Participants) | 12 | 12 | 12
mmol/L
  GSH at 0h | 1.38 (0.13) | 1.22 (0.14) | 1.23 (0.04)
  GSH at 2h | 1.12 (0.12) | 1.24 (0.07) | 1.26 (0.05)
  GSH at 4h | 1.39 (0.08) | 1.26 (0.09) | 1.30 (0.04)
  GSH at 8h | 1.40 (0.08) | 1.26 (0.08) | 1.28 (0.16)
  GSH at 24h | 1.58 (0.13) | 1.26 (0.06) | 1.31 (0.05)

2. Primary Outcome: Superoxide Dismutase (SOD) Activity in Red Blood Cells
Time Frame: 0, 2, 4, 8, 24 h
Measure: Mean (Standard Error); unit: mU/mg HgB
Arm/Group | Low Calorie Cranberry Juice Cocktail | Cranberry Leaf Extract Beverage | Non-Cranberry Beverage
Number analyzed (Participants) | 12 | 12 | 12
mU/mg HgB
  SOD at 0h | 19.0 (2.0) | 17.6 (1.0) | 20.3 (1.7)
  SOD at 2h | 19.6 (1.2) | 17.1 (1.4) | 20.7 (1.2)
  SOD at 4h | 20.9 (1.0) | 22.7 (1.4) | 19.5 (1.0)
  SOD at 8h | 16.8 (1.7) | 20.2 (1.2) | 18.2 (3.3)
  SOD at 24h | 19.2 (1.3) | 18.4 (0.7) | 14.6 (1.4)

3. Primary Outcome: Glutathione Peroxidase (GPx) Activity in Red Blood Cells
Time Frame: 0, 2, 4, 8, 24 h
Measure: Mean (Standard Error); unit: mU/mg HgB
Arm/Group | Low Calorie Cranberry Juice Cocktail | Cranberry Leaf Extract Beverage | Non-Cranberry Beverage
Number analyzed (Participants) | 12 | 12 | 12
mU/mg HgB
  GPx at 0h | 174 (14) | 161 (9) | 163 (16)
  GPx at 2h | 169 (12) | 185 (12) | 149 (14)
  GPx at 4h | 185 (14) | 197 (15) | 200 (15)
  GPx at 8h | 179 (18) | 183 (9) | 170 (29)
  GPx at 24h | 181 (15) | 172 (12) | 192 (17)

4. Primary Outcome: Oxidative Damage to DNA Assessed by Plasma 8-hydroxy-2'-Deoxyguanosine (8-OHdG)
Time Frame: 0, 2, 4, 8, 24 h
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Low Calorie Cranberry Juice Cocktail | Cranberry Leaf Extract Beverage | Non-Cranberry Beverage
Number analyzed (Participants) | 12 | 12 | 12
ng/mL
  8OHdG at 0h | 30.7 (7.9) | 33.6 (10.1) | 29.2 (6.4)
  8OHdG at 2h | 36.5 (13.3) | 31.0 (8.2) | 34.6 (9.9)
  8OHdG at 4h | 31.2 (8.8) | 33.5 (9.1) | 29.8 (6.1)
  8OHdG at 8h | 34.4 (9.7) | 31.5 (7.5) | 31.5 (9.0)
  8OHdG at 24h | 35.1 (10.5) | 32.7 (9.0) | 34.6 (10.8)

5. Primary Outcome: C-Reactive Protein (CRP) Concentrations in Plamsa
Time Frame: 0, 2, 4, 8, 24 h
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Low Calorie Cranberry Juice Cocktail | Cranberry Leaf Extract Beverage | Non-Cranberry Beverage
Number analyzed (Participants) | 12 | 12 | 12
ug/mL
  CRP at 0h | 1.10 (0.26) | 1.18 (0.34) | 0.87 (0.15)
  CRP at 2h | 0.85 (0.21) | 1.03 (0.31) | 0.99 (0.24)
  CRP at 4h | 0.69 (0.21) | 0.81 (0.20) | 0.96 (0.17)
  CRP at 8h | 1.04 (0.26) | 1.07 (0.26) | 0.99 (0.18)
  CRP at 24h | 1.28 (0.22) | 0.93 (0.20) | 0.97 (0.21)

6. Primary Outcome: Nitric Oxide (NO) Concentrations in Plamsa
Time Frame: 0, 2, 4, 8, 24 h
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Low Calorie Cranberry Juice Cocktail | Cranberry Leaf Extract Beverage | Non-Cranberry Beverage
Number analyzed (Participants) | 12 | 12 | 12
umol/L
  NO at 0h | 14.9 (1.8) | 16.6 (4.1) | 13.1 (1.4)
  NO at 2h | 13.0 (1.2) | 15.3 (3.4) | 12.2 (1.1)
  NO at 4h | 12.4 (1.2) | 10.7 (0.8) | 12.0 (1.0)
  NO at 8h | 10.5 (0.6) | 11.4 (1.3) | 10.0 (0.8)
  NO at 24h | 10.4 (0.7) | 10.6 (0.7) | 10.0 (0.5)

7. Primary Outcome: Interleukin-1alpha (IL-1a) Concentrations in Plasma
Time Frame: 0, 2, 4, 8, 24 h
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Low Calorie Cranberry Juice Cocktail | Cranberry Leaf Extract Beverage | Non-Cranberry Beverage
Number analyzed (Participants) | 12 | 12 | 12
pg/mL
  IL-1a at 0h | 17 (13) | 21 (13) | 68 (57)
  IL-1a at 2h | 49 (29) | 54 (38) | 61 (36)
  IL-1a at 4h | 30 (17) | 70 (47) | 66 (48)
  IL-1a at 8h | 43 (37) | 40 (25) | 75 (53)
  IL-1a at 24h | 33 (19) | 52 (28) | 73 (53)

8. Primary Outcome: Interleukin-1beta (IL-1b) Concentrations in Plasma
Time Frame: 0, 2, 4, 8, 24 h
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Low Calorie Cranberry Juice Cocktail | Cranberry Leaf Extract Beverage | Non-Cranberry Beverage
Number analyzed (Participants) | 12 | 12 | 12
pg/mL
  IL-1b at 0h | 22 (6) | 25 (7) | 39 (13)
  IL-1b at 2h | 35 (8) | 31 (9) | 33 (4)
  IL-1b at 4h | 26 (5) | 32 (11) | 39 (11)
  IL-1b at 8h | 24 (7) | 23 (7) | 25 (7)
  IL-1b at 24h | 26 (6) | 30 (10) | 34 (12)

9. Primary Outcome: Interleukin-2 (IL-2) Concentrations in Plasma
Time Frame: 0, 2, 4, 8, 24 h
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Low Calorie Cranberry Juice Cocktail | Cranberry Leaf Extract Beverage | Non-Cranberry Beverage
Number analyzed (Participants) | 12 | 12 | 12
pg/mL
  IL-2 at 0h | 0 (0) | 1 (1) | 13 (11)
  IL-2 at 2h | 7 (7) | 9 (9) | 6 (3)
  IL-2 at 4h | 0 (0) | 7 (6) | 5 (3)
  IL-2 at 8h | 14 (13) | 8 (7) | 10 (8)
  IL-2 at 24h | 4 (2) | 8 (6) | 13 (11)

10. Primary Outcome: Interleukin-4 (IL-4) Concentrations in Plasma
Time Frame: 0, 2, 4, 8, 24 h
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Low Calorie Cranberry Juice Cocktail | Cranberry Leaf Extract Beverage | Non-Cranberry Beverage
Number analyzed (Participants) | 12 | 12 | 12
pg/mL
  IL-4 at 0h | 15 (4) | 21 (8) | 27 (8)
  IL-4 at 2h | 19 (6) | 24 (7) | 28 (8)
  IL-4 at 4h | 13 (5) | 22 (8) | 29 (7)
  IL-4 at 8h | 15 (7) | 16 (5) | 19 (6)
  IL-4 at 24h | 16 (5) | 20 (6) | 19 (7)

11. Primary Outcome: Interleukin-6 (IL-6) Concentrations in Plasma
Time Frame: 0, 2, 4, 8, 24 h
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Low Calorie Cranberry Juice Cocktail | Cranberry Leaf Extract Beverage | Non-Cranberry Beverage
Number analyzed (Participants) | 12 | 12 | 12
pg/mL
  IL-6 at 0h | 34 (13) | 61 (36) | 74 (29)
  IL-6 at 2h | 50 (22) | 80 (34) | 56 (23)
  IL-6 at 4h | 32 (14) | 85 (51) | 61 (24)
  IL-6 at 8h | 48 (24) | 69 (31) | 68 (29)
  IL-6 at 24h | 35 (13) | 36 (16) | 62 (26)

12. Primary Outcome: Interleukin-8 (IL-8) Concentrations in Plasma
Time Frame: 0, 2, 4, 8, 24 h
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Low Calorie Cranberry Juice Cocktail | Cranberry Leaf Extract Beverage | Non-Cranberry Beverage
Number analyzed (Participants) | 12 | 12 | 12
pg/mL
  IL-8 at 0h | 7 (2) | 12 (4) | 19 (7)
  IL-8 at 2h | 11 (4) | 12 (4) | 24 (11)
  IL-8 at 4h | 8 (3) | 12 (4) | 18 (6)
  IL-8 at 8h | 11 (4) | 9 (2) | 16 (6)
  IL-8 at 24h | 11 (4) | 12 (4) | 19 (8)

13. Primary Outcome: Interleukin-10 (IL-10) Concentrations in Plasma
Time Frame: 0, 2, 4, 8, 24 h
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Low Calorie Cranberry Juice Cocktail | Cranberry Leaf Extract Beverage | Non-Cranberry Beverage
Number analyzed (Participants) | 12 | 12 | 12
pg/mL
  IL-10 at 0h | 21 (5) | 18 (5) | 19 (4)
  IL-10 at 2h | 15 (3) | 14 (4) | 14 (3)
  IL-10 at 4h | 14 (3) | 12 (4) | 14 (4)
  IL-10 at 8h | 14 (3) | 13 (4) | 17 (3)
  IL-10 at 24h | 15 (4) | 12 (4) | 14 (3)

14. Primary Outcome: Interferon-gamma (IFN-y) Concentrations in Plasma
Time Frame: 0, 2, 4, 8, 24 h
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Low Calorie Cranberry Juice Cocktail | Cranberry Leaf Extract Beverage | Non-Cranberry Beverage
Number analyzed (Participants) | 12 | 12 | 12
pg/mL
  IFN-y at 0h | 13 (7) | 20 (10) | 16 (10)
  IFN-y at 2h | 11 (6) | 17 (8) | 16 (9)
  IFN-y at 4h | 14 (8) | 16 (9) | 16 (9)
  IFN-y at 8h | 8 (6) | 14 (8) | 15 (8)
  IFN-y at 24h | 9 (6) | 10 (6) | 13 (8)

15. Primary Outcome: Tumor Necrosis Factor-alpha (TNF-a) Concentrations in Plasma
Time Frame: 0, 2, 4, 8, 24 h
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Low Calorie Cranberry Juice Cocktail | Cranberry Leaf Extract Beverage | Non-Cranberry Beverage
Number analyzed (Participants) | 12 | 12 | 12
pg/mL
  TNF-a at 0h | 23 (6) | 34 (11) | 30 (9)
  TNF-a at 2h | 24 (6) | 21 (7) | 31 (8)
  TNF-a at 4h | 20 (6) | 36 (16) | 41 (12)
  TNF-a at 8h | 18 (6) | 22 (7) | 27 (11)
  TNF-a at 24h | 19 (7) | 20 (7) | 26 (14)

16. Primary Outcome: Urinary Anti-bacteria Adhesion Activity
Time Frame: 0, 3, 6, 9, 12, 24 h
Measure: Mean (Standard Error); unit: mg PAC/mg creatinine
Arm/Group | Low Calorie Cranberry Juice Cocktail | Cranberry Leaf Extract Beverage | Non-Cranberry Beverage
Number analyzed (Participants) | 12 | 12 | 12
mg PAC/mg creatinine
  0h | 0.39 (0.14) | 0.45 (0.11) | 0.30 (0.05)
  3h | 2.34 (0.73) | 2.54 (0.61) | 1.62 (0.32)
  6h | 0.97 (0.26) | 1.05 (0.29) | 1.14 (0.37)
  9h | 0.66 (0.14) | 0.76 (0.16) | 0.59 (0.15)
  12h | 0.50 (0.07) | 0.56 (0.08) | 0.67 (0.13)
  24h | 0.38 (0.06) | 0.48 (0.07) | 0.54 (0.10)

ADVERSE EVENTS:
Arm/Group | Low Calorie Cranberry Juice Cocktail | Cranberry Leaf Extract Beverage | Non-Cranberry Beverage
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No